CLINICAL TRIAL: NCT02901301
Title: A Phase Ib/II Study of First Line Pembrolizumab in Combination With Trastuzumab, Capecitabine, and Cisplatin in HER2 Positive Gastric Cancer
Brief Title: Pembrolizumab, Trastuzumab, HER2 Positive Gastric Cancer
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Principal Investigator, Hyun Cheol Chung, Professor, Yonsei University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4-2016-0190
Record Dates: First submitted 2016-09-11; First posted 2016-09-15 (Estimated); Last update posted 2021-04-06 (Actual); Status verified 2021-04

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — pembrolizumab; Trastuzumab; Capecitabine; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 4 combination (Experimental): pembrolizumab 200mg, IV, q3weeks, Day 1 trastuzumab 6mg/kg (8mg loading dose), IV, q3weeks, Day 1 capecitabine 1000mg/m2, PO, BID, Day 1-14 cisplatin 80mg/m2 (level 1), IV, q3weeks, Day 1
  Interventions: Drug: Pembrolizumab; Drug: Trastuzumab; Drug: Capecitabine; Drug: Cisplatin

INTERVENTIONS:
Drug: Pembrolizumab — 200mg, IV, q3weeks, Day 1
Drug: Trastuzumab — 6mg/kg (8mg loading dose), IV, q3weeks, Day 1
Drug: Capecitabine — 1000mg/m2, PO, BID, Day 1-14
Drug: Cisplatin — 80mg/m2 (level 1), IV, q3weeks, Day 1

SUMMARY:
Gastric cancer is one of the major health problems worldwide, and one of the leading cause of death especially in Asia. Though the cytotoxic chemotherapy is the main treatment option, newer and molecularly targeted agents are recently incorporated to improve the survival outcome. Human epidermal growth factor receptor 2 (HER2, ErbB2) is a transmembrane tyrosine kinase receptor and is overexpressed or amplified in 10-20% of gastric cancer. Recently, Trastuzumab for Gastric Cancer (ToGA) study reported the clinical benefit of trastuzumab for HER2 positive gastric cancer patients. However, because the majority of patients develop intrinsic or acquired resistance within 1 year, elucidating the molecular mechanisms for trastuzumab resistance is warranted to improve the survival outcome of HER2 positive gastric cancer patients.

A growing body of preclinical and clinical evidence shows that the immune system contributes substantially to the therapeutic effects of "monoclonal antibody, trastuzumab" in solid tumors. Pembrolizumab is a potent and highly selective humanized monoclonal antibody designed to directly block the interaction between PD-1 and its ligands, PD-L1 and PD-L2.

Based on strong rationale in exploring the impact of combining trastuzumab with anti-PD-1 inhibitor in HER2 positive cancer, we suggest multicenter phase IB/II study to determine antitumor activity and safety of pembrolizumab in combination with standard treatment (trastuzumab, capecitabine, and cisplatin) in patients with HER2 positive gastric cancer.

ELIGIBILITY:
Inclusion Criteria:

1. HER2 positive advanced gastric cancer
2. Be willing and able to provide written informed consent/assent for the trial.
3. Be 19 years of age on day of signing informed consent.
4. Have measurable disease based on RECIST 1.1.
5. performance status of 0 or 1 on the Eastern Cooperative Oncology Group Performance Scale.
6. Demonstrate adequate organ function
7. Female subject of childbearing potential should have a negative urine or serum pregnancy or be willing to use birth control.

Exclusion Criteria:

1. Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of treatment.
2. Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment.
3. Has a known history of active Bacillus Tuberculosis
4. Hypersensitivity to pembrolizumab or any of its excipients.
5. Has had a prior anti-cancer monoclonal antibody within 4 weeks prior to study Day 1 or who has not recovered from adverse events due to agents administered more than 4 weeks earlier.
6. Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study Day 1 or who has not recovered from adverse events due to a previously administered agent.
7. Has a known additional malignancy that is progressing or requires active treatment within 3 years.
8. Has known active central nervous system metastases and/or carcinomatous meningitis.
9. Has active autoimmune disease that has required systemic treatment in the past 2 years
10. Has known history of, or any evidence of active, non-infectious pneumonitis.
11. Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent.
12. Has known active Hepatitis B or Hepatitis C
13. Has received a live vaccine within 30 days of planned start of study therapy.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2017-02-06 (Actual); Primary Completion 2020-10-31 (Actual); Study Completion 2021-10 (Estimated)

PRIMARY OUTCOMES:
The recommended dose of phase II | 4 weeks
The overall response rate using RECIST 1.1 | 6 weeks

SECONDARY OUTCOMES:
Duration of response | 1 year
Time to response | 6 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Yonsei University Health System, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Jung SH, Lee CK, Kwon WS, Yun S, Jung M, Kim HS, Chung HC, Chung YJ, Rha SY. Monitoring the Outcomes of Systemic Chemotherapy Including Immune Checkpoint Inhibitor for HER2-Positive Metastatic Gastric Cancer by Liquid Biopsy. Yonsei Med J. 2023 Sep;64(9):531-540. doi: 10.3349/ymj.2023.0096. PMID 37634629
- [Derived] Lee CK, Rha SY, Kim HS, Jung M, Kang B, Che J, Kwon WS, Park S, Bae WK, Koo DH, Shin SJ, Kim H, Jeung HC, Zang DY, Lee SK, Nam CM, Chung HC. A single arm phase Ib/II trial of first-line pembrolizumab, trastuzumab and chemotherapy for advanced HER2-positive gastric cancer. Nat Commun. 2022 Oct 12;13(1):6002. doi: 10.1038/s41467-022-33267-z. PMID 36224176